CLINICAL TRIAL: NCT03698838
Title: A Pilot, Prospective Study of Myelin Imaging Changes in Patients With Neurosurgical Diseases
Brief Title: Myelin Imaging Changes In Patients With Neurosurgical Diseases
Acronym: McDESPOT
Status: Terminated | Type: Observational
Why Stopped: Principal Investigator left Institution
Sponsor: Memorial Healthcare System (Other)
Responsible Party: Sponsor
Other Study IDs: McDESPOT
Record Dates: First submitted 2018-10-04; First posted 2018-10-09 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Hydrocephalus in Children; Epilepsy; Craniosynostoses; Traumatic Brain Injury
MeSH Terms: conditions — Epilepsy; Craniosynostoses; Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- McDESPOT Study Group: Patients aged 0-19 who have an MRI ordered clinically and have one of the following conditions: epilepsy, hydrocephalus, craniosynostosis or mild traumatic brain injury. Epilepsy, hydrocephalus and craniosynostosis patients will be both newly diagnosed and chronic. MTBI patients will be acute and chronic and defined as a glascow coma score (GCS) of 13-15.These patients will have a 10 minute MRI sequence (McDESPOT) added to their standard of care T1 and T2 scans.
  Interventions: Device: McDESPOT
- Control Model: Control model derived from a linear mixed-effects model (Spader et al 2013)

INTERVENTIONS:
Device: McDESPOT — MRI sequence, mcDESPOT (multicomponent driven equilibrium potential of T1 and T2) that utilizes a computer model that takes T1 and T2 sequences and derives a quantitative value for the myelin content in the myelin sheath
  Groups: McDESPOT Study Group

SUMMARY:
Investigate myelin alterations in patients with neurosurgical diseases

DETAILED DESCRIPTION:
While a number of advanced imaging techniques, notably magnetization transfer, diffusion tensor and quantitative T1 and T2 imaging (MTI, DTI, qT1 and qT2, respectively), have been used previously to study white matter in neurosurgical diseases, these methods provide only indirect, non-specific information related to myelin content. For example, these modalities can tell when there is swelling that is affecting the movement of water, which may be indicative of a process that would affect myelin, but they cannot tell us specific information about the amount of myelin surrounding a nerve.

The investigators propose using a MRI sequence, mcDESPOT (multicomponent driven equilibrium potential of T1 and T2) that utilizes a computer model that takes T1 and T2 sequences and derives a quantitative value for the myelin content in the myelin sheath.

In the present program, the investigators propose adding the mcDESPOT sequence to the MRI scanner in accordance with the MRI manufacturer's technical requirements. When this sequence is added, the normal sequences are done first and mcDESPOT is done last. Although the sequences obtained for mcDESPOT are sequences used in clinical practice, the flip-angles are changed so that they cannot be read like a traditional image. Rather, the data have to be post-processed by a computer in order to be able to derive myelin information.

McDESPOT is a 10 minute sequence that can be added to any MRI scanner. It is a obtained from standard T1 and T2 sequences.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age range: 0-19
2. Patients who have an MRI ordered clinically and have one of the following conditions: epilepsy, hydrocephalus, craniosynostosis or mild traumatic brain injury. Epilepsy, hydrocephalus and craniosynostosis patients will be both newly diagnosed and chronic. MTBI patients will be acute and chronic and defined as a glascow coma score (GCS) of 13-15.
3. Patients or their proxy should be capable of giving informed consent

Exclusion Criteria:

1. Unable to tolerate an extra 10 minutes of MRI scan

Max Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients aged 0-19 who have an MRI ordered clinically and have one of the following conditions: epilepsy, hydrocephalus, craniosynostosis or mild traumatic brain injury. Epilepsy, hydrocephalus and craniosynostosis patients will be both newly diagnosed and chronic. MTBI patients will be acute and chronic and defined as a glascow coma score (GCS) of 13-15.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
Myelin Alterations Read on MRI sequence | 10 minutes
  Investigate myelin alterations in patients with neurosurgical diseases with McDESPOT sequence on MRI scanner for T1 and T 2 scans.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Spader, MD, Principal Investigator — Memorial Healthcare System
Locations (1):
- Memorial Healthcare System, Hollywood, Florida, United States

IPD SHARING:
Plan to Share IPD: No